CLINICAL TRIAL: NCT06514261
Title: Phase 1 Trial of Iadademstat in Combination With Venetoclax and Azacitidine in Patients With Treatment Naive AML
Brief Title: Testing the Combination of an Anti-Cancer Drug, Iadademstat, With Other Anti-Cancer Drugs (Venetoclax and Azacitidine) for Treating AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-04616; NCI-2024-04616 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-115; 10630 (Other: UPMC Hillman Cancer Center LAO); 10630 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2024-07-20; First posted 2024-07-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Specimen Handling; iadademstat; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (iadademstat, venetoclax, azacitidine) (Experimental): INDUCTION: Patients receive iadademstat PO QD on days 1-5, 8-12, and may also receive it on days 15-19 of each cycle, venetoclax PO QD on days 1-14 or 1-21 of each cycle, and azacitidine IV over 10-40 minutes or SC on days 1-7 of each cycle or days 1-5 and 8-9 after cycle 1. Cycles repeat every 28 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may also undergo buccal swab collection on study.
  CONSOLIDATION: Patients receive iadademstat PO QD on days 1-5, 8-12 and may also receive it on days 15-19 of each cycle, venetoclax PO QD on days 1-7 or 1-14 of each cycle, and azacitidine IV over 10-40 minutes or SC on days 1-7 of each cycle or days 1-5 and 8-9 after cycle 1. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection and may undergo bone marrow aspiration throughout the study.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Buccal Swab; Drug: Iadademstat; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Buccal Swab — Undergo buccal swab
  Other Names: Buccal Scraping; Buccal Smear; Buccal swab/scraping; Buccal Swabbing
Drug: Iadademstat — Given PO
  Other Names: ORY 1001; ORY-1001; RG 6016; RG6016; RO 7051790; RO7051790; trans-N1-((1R,2S)-2-Phenylcyclopropyl)-1,4-cyclohexanediamine
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I trial tests safety, side effects and best dose of iadademstat with azacitidine and venetoclax for the treatment of patients with acute myeloid leukemia (AML) who have not received treatment (treatment naive). Chemotherapy drugs, such as iadademstat and azacitidine work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving iadademstat with azacitidine and venetoclax may be safe and tolerable in treating patients with treatment naive AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase 2 dose (RP2D) and safety profile of iadademstat in combination with venetoclax and azacitidine.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity, including evaluating the overall response rate (ORR), defined as complete remission (CR), CR with incomplete hematologic recovery (Cri), or CR with partial hematologic recovery (CRh).

II. To evaluate the measurable residual disease (MRD)-negative composite CR (cCR) rate after 1, 2, and 3 cycles using multiparameter flow cytometry (MFC) and evaluate event-free survival (EFS), overall survival (OS), and duration of response (DoR).

III. To determine if treatment will be associated with expansion of high risk molecular (PTPN11, NRAS, KRAS, NF1, and TP53) and cytogenetic (complex karyotype) markers over time.

EXPLORATORY OBJECTIVES:

I. To determine the rate of MRD-negative cCR across molecular (PTPN11, NRAS, KRAS, NF1, and TP53) and cytogenetic (complex karyotype) subgroups.

II. To document the effect of therapy on LSD1-target engagement.

III. To determine if secondary resistance (remission with therapy then relapse) in both arms is associated with:

IIIa. Acquisition of resistance mutations including BCL-2 and BAX; IIIb. Development or expansion of mutations that activate RAS/MAPK/FLT3 including NRAS, KRAS, PTPN11, NF1, and FLT3-ITD; IIIc. Over-expression of resistance proteins such as MCL-1 or BCL-XL. IV. To determine pharmacokinetics (PK) in the triplet therapy of iadademstat, azacitidine, and venetoclax.

V. To explore PK/pharmacodynamic (PD) relationship of iadademstat and venetoclax in patients who received the triplet therapy of iadademstat, azacitidine, and venetoclax.

VI. To evaluate the association between time to achieve an MRD-negative cCR and EFS, OS, and DoR.

OUTLINE: This is a dose-escalation study of iadademstat and venetoclax in combination with azacitidine.

INDUCTION: Patients receive iadademstat orally (PO) once daily (QD) on days 1-5, 8-12, and may also receive it on days 15-19 of each cycle, venetoclax PO QD on days 1-14 or 1-21 of each cycle, and azacitidine intravenously (IV) over 10-40 minutes or subcutaneously (SC) on days 1-7 of each cycle or days 1-5 and 8-9 after cycle 1. Cycles repeat every 28 days for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients may also undergo buccal swab collection on study.

CONSOLIDATION: Patients receive iadademstat PO QD on days 1-5, 8-12 and may also receive it on days 15-19 of each cycle, venetoclax PO QD on days 1-7 or 1-14 of each cycle, and azacitidine IV over 10-40 minutes or SC on days 1-7 of each cycle or days 1-5 and 8-9 after cycle 1. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection and may undergo bone marrow aspiration throughout the study.

After completion of study treatment, patients are followed every 3-4 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have established and confirmed diagnosis of intermediate or adverse-risk AML according to the European LeukemiaNet 2022 classification criteria
* Previously untreated AML excluding hydroxyurea and all-trans retinoic acid (ATRA). ATRA would only be used for suspected AML
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of iadademstat in combination with venetoclax and azacitidine in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Patient is able to swallow oral medications
* Patient must have a body weight of at least 50 kg due to the use of flat doses
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) OR direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 x ULN or ≤ 3 x ULN if patient has Gilbert's disease
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 × institutional ULN or < 5 ULN if due to AML
* Chronic kidney disease (CKD)-epidemiology collaboration (EPI) glomerular filtration rate (GFR) ≥ 40 mL/min/1.73 m^2
* Peripheral white blood cell (WBC) count < 25 x 10^9/L on day 1 prior to treatment initiation. Hydroxyurea for up to 2 weeks is allowed for cytoreduction until 24 hours prior to study treatment
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better. Patients with a troponin leak (i.e. elevated troponin levels at presentation without evidence of an active myocardial infarction (MI) are eligible
* The effects of iadademstat on the developing human fetus are unknown. For this reason and because LSD1 inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, females of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 180 days after the last dose of study medication. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Males with female partners of child-bearing potential treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 180 days after the last dose of study medication. Women of child-bearing potential agree not to donate or freeze egg(s) during the course of this study or within 180 days after receiving their last dose of study drug. Male patients agree not to donate sperm during the course of this study or within 180 days after receiving their last dose of study drug
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients are willing and able to receive intensive induction chemotherapy
* Patients have isolated myeloid sarcoma or acute promyelocytic leukemia (APL) French-American-British (FAB) M3
* Patients who have not recovered from adverse events of grade 3 or more due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* Patients who have active central nervous system (CNS) involvement by AML
* Patients who have disseminated intravascular coagulopathy with active systemic bleeding or venous or atrial signs of thrombosis
* Patients who require treatment while on study with concomitant drugs that target the 5HT2B receptor or the sigma nonspecific receptor (e.g., escitalopram, fluoxetine, sertraline) except for drugs that are considered absolutely essential for the care of the patient and with appropriate treatment monitoring
* Patients with manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of oral drugs. In addition, patients with enteric stomata are also excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to iadademstat, azacitidine, mannitol, or venetoclax
* Iadademstat Concomitant Medication Considerations: Patients are not allowed to receive prophylactic hematopoietic colony stimulating factors, any complementary or alternative medicine (any of various systems of healing or treating disease [as non-prescription drugs, herbal medicine and homeopathy])
* Patients should not use strong CYP3A inhibitors with the exception of antifungals for which standard of care (SOC) dose modifications of venetoclax exist
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous. This includes, but is not limited to:

  * Myocardial infarction with evidence of residual abnormalities within 3 months prior to enrollment (Troponin leak alone not included if no residual dysfunction);
  * New York Heart Association (NYHA) Class III or IV heart failure;
  * Severe uncontrolled ventricular arrhythmias;
  * Electrocardiographic evidence of acute ischemia or active life-threatening conduction system abnormalities:

    * Since patients with AML frequently require supportive care with agents that affect the corrected QT interval (QTc), if clinically indicated, obtain an electrocardiogram (ECG) prior to enrollment
* As infection is a common feature of AML, patients with active infection are permitted to enroll provided that the infection is under control (i.e., no signs of severe systemic inflammatory response that makes patient clinically unstable in the opinion of the investigator, and the patient is hemodynamically stable). Patients with uncontrolled infection shall not be enrolled until the infection is treated and brought under control
* Pregnant women are excluded from this study because iadademstat is LSD1 inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with iadademstat, breastfeeding should be discontinued if the mother is treated with iadademstat. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | Up to completion of cycle 1
  DLT is defined as any of the following treatment emergent adverse events occurring in the first cycle that are related (possibly, probably, or definitely) to administration of the study agents. Will utilize National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 for toxicity grading and reporting.
Incidence of adverse events (AEs) | Up to completion of therapy
  Will utilize NCI-CTCAE v5.0 for AE grading and reporting.

SECONDARY OUTCOMES:
Objective response rate | Up to 4 years
  The probability of achieving a complete remission (CR), CR with incomplete hematologic recovery (CRi), CR with partial hematologic recovery (CRh), will be estimated with exact 95% binomial confidence intervals.
Morphologic leukemia free state | Up to 4 years
Minimal residual disease (MRD)-negative composite complete remission (cCR) | After completion of 2 cycles
  Will be estimated with exact 95% binomial confidence intervals.
Event free survival | From study enrollment to disease progression, treatment failure (failure to achieve CR or < 5% bone marrow blasts) confirmed relapse or death, up to 4 years
  Will be estimated by the Kaplan-Meier method, along with 95% confidence regions.
Overall survival | Up to 4 years
  Will be estimated by the Kaplan-Meier method, along with 95% confidence regions.
Duration of response | Up to 4 years
  Will be estimated by the Kaplan-Meier method, along with 95% confidence regions.
Proportion of patients with high risk molecular and cytogenetic markers | At baseline, during treatment, and at progression of disease, up to 4 years
  Will be estimated with exact 95% binomial confidence intervals and compared between baseline, during treatment, and at progression of disease.

OTHER OUTCOMES:
MRD-negative cCR and molecular/cytogenetic risk group status | After cycles 1, 3 and 6
  Rates of MRD-negative cCR will be tabulated descriptively across molecular (PTPN11, NRAS, KRAS, NF1, and TP53) and cytogenetic (complex karyotype) subgroups. Will be estimated with exact 95% binomial confidence intervals.
Percentage LSD1 target engagement by chemoprobe in peripheral blood mononuclear cells | Up to 4 years
  Changes in %LSD1 target engagement will be compared between patients and between dose levels to confirm target engagement. Data between dose levels will be compared with a rank sum test and within patients with a signed rank test and/or mixed effects regression. Data between dose levels will be compared with a rank sum test and within patients with a signed rank test and/or mixed effects regression.
BCL-2 mutations by next generations sequencing (NGS) in bone marrow (BM) of patients who initially respond and then progress | At baseline, during treatment, and at progression of disease, up to 4 years
BAX mutations by NGS in BM of patients who initially respond and then progress | At baseline, during treatment, and at progression of disease, up to 4 years
Mutations by NGS in relevant genes in BM of patients who initially respond and then progress | At baseline and at progression of disease, up to 4 years
Expression of MCL-1, BCL-XL and related proteins in PBMCs of patients who initially respond and then progress | At baseline, during treatment, and at progression of disease, up to 4 years
Venetoclax trough | Day 5, 8 and 12
Iadademstat trough and derived pharmacokinetic parameters | Up to 4 years
Event free survival | From study enrollment to disease progression, treatment failure (failure to achieve CR or < 5% bone marrow blasts) confirmed relapse or death, up to 4 years
  Kaplan Meier methods will be used to estimate the median survivals (with a 90% confidence interval) as a function of time to response. The effects of time to response will also be tested with a Cox proportional hazard model, after controlling for risk factors or confounders. In addition, will evaluate EFS within the subpopulation of patients that started continued treatment.
Overall survival | Up to 4 years
  Kaplan Meier methods will be used to estimate the median survivals (with a 90% confidence interval) as a function of time to response. The effects of time to response will also be tested with a Cox proportional hazard model, after controlling for risk factors or confounders. In addition, will evaluate OS within the subpopulation of patients that started continued treatment.
Duration of response | Up to 4 years
  Kaplan Meier methods will be used to estimate the median survivals (with a 90% confidence interval) as a function of time to response. The effects of time to response will also be tested with a Cox proportional hazard model, after controlling for risk factors or confounders. In addition, will evaluate duration of response within the subpopulation of patients that started continued treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Annie P Im, Principal Investigator — University of Pittsburgh Cancer Institute LAO
Locations (4):
- United States (4):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm